CLINICAL TRIAL: NCT05366387
Title: Effect of Intrapulmonary Percussion Ventilation on Deposition of Inhaled Aerosols in Idiopathic Pulmonary Fibrosis
Acronym: AEROPERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DR210241; 2021-A02003-38 (Other: IdRCB); 22.00149.000065 (Other: CPP (SI RIPH 2G))
Record Dates: First submitted 2022-03-25; First posted 2022-05-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: aerosol; deposition; Intrapulmonary Percussive Ventilation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Phase 1 : Delivery of intrapulmonary percussive ventilation (IPV) to assess for discomfort and adverse effects Phase 2 : Delivery of radiolabelled aerosols with or without IPV, in a crossover design
Who Masked: Outcomes Assessor
Masking Description: Phase 1 : Open label Phase 2 : The primary endpoint is defined by quantitative analysis of SPECT images. Analysis is done by a project Partner (Inserm UMR1101), blinded to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerosol delivery without intrapulmonary percussive ventilation (Control condition) (Sham Comparator): A radiolabelled 99mTc-DTPA aerosol is generated with a jet nebuliser and is inhaled by the subject through a device (connecting tubes, filters) connecting the nebuliser with 1) a mouthpiece and 2) an intrapulmonary percussive ventilation device which is turned off.
  Aerosol deposition in fibrotic lung regions is characterized by SPECT imaging.
  Interventions: Radiation: delivery of 99mTc-DTPA aerosol
- Aerosol delivery with intrapulmonary percussive ventilation (IPV condition) (Active Comparator): A radiolabelled 99mTc-DTPA aerosol is generated with a jet nebuliser and is inhaled by the subject through a device (connecting tubes, filters) connecting the nebuliser with 1) a mouthpiece and 2) an intrapulmonary percussive ventilation device which is turned on (frequency=1 Hz, pressure to be determined in phase 1 for each patient, in the 5-40 cm H2O range).
  Aerosol deposition in fibrotic lung regions is characterized by SPECT imaging.
  Interventions: Device: intrapulmonary percussive ventilation; Radiation: delivery of 99mTc-DTPA aerosol

INTERVENTIONS:
Device: intrapulmonary percussive ventilation — Intrapulmonary percussive ventilation is a non invasive ventilation technique where small boli or air are delivered, at adjustable frequency and pressure, to the upper airways though a mouthpiece. IPV is currently used in the clinic to aid with airway clearance in neuromuscular and airway diseases.
  Arms: Aerosol delivery with intrapulmonary percussive ventilation (IPV condition)
Radiation: delivery of 99mTc-DTPA aerosol — A 99mTc-DTPA aerosol (500 MBq+/-20%, 3 ml volume) is generated with a jet nebuliser (MMAD 4 µm). The aerosol is inhaled by the study subject and lung deposition is imaged by SPECT

SUMMARY:
This protocol aims to evaluate the feasibility and benefit of Intrapulmonary Percussive Ventilation (IPV) to improve deposition of inhaled radiolabelled aerosols in fibrotic lung regions of patients with Idiopathic Pulmonary Fibrosis (IPF).

Phase 1 of the protocol aims to identify the highest IPV pressure that is tolerated by individual patients. Secondary endpoints explore safety of IPV in IPF patients.

Phase 2 of the protocol is a crossover randomized trial where patients will inhale 99mTc-labelled DiethyleneTriamine PentaAcetate (DTPA) aerosols with or without IPV. Aerosol deposition in HRCT-defined fibrotic regions of interest (ROI) is described by Single Photon Emission Computed Tomography (SPECT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF according to 2018 ATS/ERS/JRS/ALAT guidelines
* Affiliation to health insurance
* Signed informed consent

Exclusion Criteria:

* Other chronic lung disease
* Airflow obstruction (FEV1/FVC<0.7)
* History of congestive heart failure
* History of IPF exacerbation
* History of lung cancer
* Chronic cough precluding aerosol delivery and radioprotection
* Claustrophobia
* 24h/24 oxygen therapy
* Any acute lung disease
* Any potentially transmissible lung infection
* Current or possible pregnancy and breastfeeding
* Contra-indications to IPV : Emphysema, recent barotrauma, pneumothorax, pneumomediastinum
* History of pneumothorax or pneumomediastinum
* Patient unable to hold a mouthpiece tightly
* Patient under legal protection (guardianship, curatorship)
* Contraindication to the administration of Technescan DTPA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Phase 1: Discomfort during IPV | immediately after IPV (visit V1)
  IPV is delivered at increasing pressure (from 5 cm H2O to 40 cm H2O maximum pressure) and discomfort is assessed by a 5-level Likert scale ranging from "no discomfort" to "untolerable discomfort". IPV is stopped when discomfort is rated as "difficult to tolerate" whatever the pressure.
Phase 2: Change between Control and IPV condition in amount of 99mTc-labelled DTPA aerosol deposited in fibrotic lung regions, reported to loaded dose | After delivery of radiolabelled aerosol under both Control and IPV condition (Visit 4/5) i.e. up to 1 month
  Following aerosol delivery, chest imaging is done with a SPECT device. SPECT images are fused to high resolution computed tomography (HRCT) images. Fibrotic lung regions regions of interest (ROI) are defined by analysis of HRCT images.
  SPECT signal in fibrotic ROI is reported to the radioactive dose that was loaded in the nebulizer
  Endpoint is radioactive signal in fibrotic ROI / loaded dose

SECONDARY OUTCOMES:
Phase 1: Sensations associated with IPV in patients with IPF | immediately after IPV (Visit 1)
  5-levels Likert scales ranging from "not at all" to "Very much" are used to answer the following questions : "I have trouble breathing" "This thumps to much" "This is scary"
Phase 1: IPV-induced variations in dyspnea | Before IPV (Visit 1) and 15 days after IPV (Visit 2)
  Dyspnea-12 scale
Phase 1: IPV-induced variations in cough | Before IPV (Visit 1) and 15 days after IPV (Visit 2)
  Leicester Cough Questionnaire
Phase 1: IPV-induced variations in Forced Vital Capacity | Before IPV (Visit 1) and 15 days after IPV (Visit 2)
  Spirometry Forced vital capacity is expressed in liters
Phase 1: IPV-induced variations in Carbon monoxide transfer factor (DLCO) | Before IPV (Visit 1) and 15 days after IPV (Visit 2)
  Single breath test DLCO is expressed in mL/min/mmHg
Phase 1: IPV-induced variations in 5 Hz respiratory reactance | Before IPV (Visit 1) and 15 days after IPV (Visit 2)
  Impulse oscillometry 5 Hz reactance is expressed as kPa.s/L
Phase 1: Incidence of Treatment-Emergent Adverse Events | immediately after IPV (Visit 1) until 15 days after IPV (V2)
  Symptomatic pneumothorax Acute exacerbation of IPF requiring hospitalization
Phase 2 : Change between Control and IPV condition in total lung deposition of the 99mTc-labelled DTPA aerosol | After delivery of radiolabelled aerosol under both Control and IPV condition (Visit 5)
  Ratio of SPECT in total lung / loaded dose
Phase 2: Ratio of deposition of the 99mTc-labelled DTPA aerosol in fibrotic lung versus normal lung | After aerosol delivery in the Control condition
  ROI for normally-appearing lung are defined by HRCT. Endpoint is SPECT signal in fibrotic lung ROI / SPECT signal in normally-appearing lung ROI
Incidence of Treatment-Emergent Adverse Events one month after treatment | 1-month after the last aerosol delivery (V6)
  Telephone interview to assess for :
  Symptomatic pneumothorax Acute exacerbation of IPF requiring hospitalization

OTHER OUTCOMES:
Exploratory endpoint : Impact of specific lung lesions on pulmonary ventilation and deposition of the 99mTc-labelled DTPA aerosol | After aerosol delivery under the Control condition (Visit 4 or 5 according to randomization) i.e. up to 1 month
  Additional ROI are defined on HRCT to define predominant lung lesions as either "ground glass opacities", "reticulations", or "bronchiectasis".
  The impact of these lesions on pulmonary ventilation and aerosol deposition is described as :
  * pulmonary ventilation : Fusion of HRCT images with 88mKr-ventilation SPECT images.
  * aerosol deposition : Fusion of HRCT images with 99mTc-DTPA aerosol deposition images.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PLANTIER, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Pulmonology Department, University Hospital, Tours, Tours, France